CLINICAL TRIAL: NCT04248777
Title: LEft Main Oct Guided iNterventions
Brief Title: Optical Coherence Tomography - Guided Protocol for Left Main Percutaneous Coronary Intervention
Acronym: LEMON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Mutualiste Montsouris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CARDIO-2017-01
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Left Main Coronary Artery Stenosis
Keywords: Optical Coherence Tomography (OCT); Percutaneous Coronary Intervention (PCI).

STUDY DESIGN:
Intervention Model Description: Patients with left main artery planned PCI for stable or unstable coronary artery disease.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- left main PCI guided by OCT (Other): The LM PCI strategy is guided by 3 OCT runs, according to a pre-defined standardized protocol.
  Interventions: Other: standardised OCT-guided intervention

INTERVENTIONS:
Other: standardised OCT-guided intervention — The first OCT run (run1) analyse plaque characteristics, identify proximal and distal landing zones (according to previously published criteria) , measure lesion length and reference segments dimensions (diameters and luminal areas). The second run (run2) aims to assess adequate guidewire recrossing point into stent jailed side branch and identify early stent mechanical non-optimal results. The third run (run3) analyse final stent expansion and identify major struts malposition and edge dissection.

SUMMARY:
LEMON aim is to evaluate the feasibility, efficiency and security of a standardized Optical Coherence Tomography (OCT) - guided protocol for completion and optimization of Left Main (LM) Percutaneous Coronary Intervention (PCI).

DETAILED DESCRIPTION:
The LEMON study (LEft Main Oct-guided iNterventions) is a prospective, multicentre, open-label, interventional , non-randomized trial that investigates the feasibility and efficiency of OCT guidance for left main PCI in 10 active French interventional cardiology centres. The aim of the study is the appliance of a pre-defined standardized protocol for LM PCI . The LM PCI strategy is guided by 3 OCT runs, according to a pre-determined protocol. The first OCT run (run1) is performed before any stent implantation, the second run (run2) is performed after the stent is implanted, POT (proximal optimization technique) is applied and side branch iss rewired through stent struts. The third run (run3) is performed after PCI optimization. In case of additional stent optimization, a supplementary OCT run is applied in order to assess final result.

ELIGIBILITY:
Inclusion Criteria:

* age >18
* stable or non-stable distal Left Main lesion (with or without previous Coronary Artery Bypass Graft), involving or not Left Anterior Descending and Coronary Circumflex ostias and requiring Percutaneous Coronary Intervention with a one or two stents strategy
* stable or non-stable ostial Left Anterior Descending and/or Coronary Circumflex lesion requiring Percutaneous Coronary Intervention with involvement of distal Left Main
* SYNTAX angiographic score <23
* informed consent

Exclusion Criteria:

* ostial Left Main lesion
* on-going acute STEMI
* on-going cardiogenic shock
* severe chronic renal failure (Cr Cl <30 ml/min/m2)
* anticipated technical contra-indication to OCT (highly calcified lesions, severe proximal tortuosity)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
success of the OCT procedure | Post PCI / Immediate
  score Thrombolysis In Myocardial Infarction (TIMI) equal to 3 in all vessels, 50% residual stenosis in the various angiography segments, adequate expansion according to minimum intra stent area > 80% of the luminal area of the reference segment on Main Vessel and Main Branch.

SECONDARY OUTCOMES:
incidence of major adverse cardiovascular events | 30 days post PCI
  death, cardiovascular death, stent thrombosis, target vessel revascularization
rate of appropriate wire position | 30 days post PCI
  percentage of appropriate wire position in adequate stent cell before side branch ostium dilation.
rate of appropriate stent expansion according to DOCTORS and ILUMIEN-III criteria. | 30 days post PCI
  percentage of stent expansion according to DOCTORS and ILUMIEN-III

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas AMABILE, MD,PhD, Principal Investigator — Institut Mutualiste Montsouris
Locations (11):
- France (11):
  - Chu Besancon, Besançon
  - Chu Bordeaux, Bordeaux
  - Clinique Saint Augustin, Bordeaux
  - Hôpital privé Saint Martin, Caen
  - Chu Clermont Ferrand, Clermont-Ferrand
  - Ch Chartres, Le Coudray
  - Institut hospitalier Jacques Cartier, Massy
  - Ch Annecy Genevois, Metz-Tessy
  - CHU Nîmes, Nîmes
  - Institut Mutualiste Montsouris, Paris
  - Clinique Saint Hilaire, Rouen

IPD SHARING:
Plan to Share IPD: No